CLINICAL TRIAL: NCT05175365
Title: Dance in Parkinson's Disease: An Optimized and Adapted Approach to Promote the Well-being and Functional Status of Patients
Brief Title: The Impact of Dancing in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Kinésiphilia (Unknown)
Responsible Party: Principal Investigator, Helena Cassol, Principal Investigator, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-313
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance (Experimental): Patients allocated to this group will attend dance classes for patients with Parkinson's disease given once a week over a 4-month period for a total of 16 dance sessions.
  Interventions: Behavioral: Dance
- Control (No Intervention): The control group will receive its rehabilitation care.

INTERVENTIONS:
Behavioral: Dance — Each session consists of a 60-minute dance class taught by a professional dancer. Dance classes begin with a seated warm-up with various coordination, rhythm, range of motion, memorization and coordination exercises. The level of difficulty of the exercises increases as the sessions progress. Balance is also an important part of training as well as the feeling of being part of a group, of interacting with each other. The hour ends with stretching in a sitting position.
  Arms: Dance

SUMMARY:
This clinical study intends to confirm the results of previous studies showing the positive effect of dance on patients with Parkinson's disease on both mental and physical health via a randomized controlled trial. Patients will be randomized into the intervention group (dance courses in addition to standard care) or in the control group (standard care).

DETAILED DESCRIPTION:
This is a clinical study on the benefits of dance in Parkinson's disease. In recent years, dance has become an interesting strategy to promote motor and non-motor functions in Parkinson's disease. More than a rehabilitation strategy, dance appears to be an optimal approach to promote functional outcomes as it combines physical, rhythmic, cognitive, emotional and social elements that could have a positive impact on multiple impairments in Parkinson's disease. The investigators believe that the notion of pleasure is crucial for rehabilitation, especially in people suffering from depression, and that it is often not taken into account in conventional rehabilitation strategies.

The goal of the present study is to confirm these preliminary results. This clinical study will run over two years, from January 2022 to January 2024, but an experimental session will last 4 months. The aim of this protocol is to better characterize the impact of dance on well-being, disease progression and possible neuronal reorganization in patients with Parkinson's disease. A better quality of life, a higher level of satisfaction and an improvement in functional status are expected in the experimental group.

During this study, three examinations will be carried out over 4 months. One at the start of the study, one at mid-term (after 8 weeks) and one at the end of the study. These evaluations will take place at the place of the dance lessons for the experimental group and within the university hospital for the control group.

Assessment will be done through different scales and questionnaires to assess well-being, satisfaction, feelings of happiness, functional status, cognitive functions and the correlation between functional and cognitive progress and neuronal activity.

This study is a "controlled and randomized" study that is to say that in a random manner, half of the participants will participate in weekly dance sessions lasting 60 minutes in addition to their conventional physiotherapy sessions while the control group will only receive conventional physiotherapy sessions during the first 4 months but will still benefit from dance sessions after the 4 months of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's disease
* Hoehn & Yahr Stadium <3
* Signature of the written consent form

Exclusion Criteria:

* No cardiac or respiratory or neurological or rheumatological disease incompatible with the practice of a physical activity
* Has not had any surgery interfering with motor function in the past 6 months
* Has no cognitive impairment - MoCA <26
* Does not present hearing problems that do not all

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire (PDQ-39) | 16 weeks
  This questionnaire assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. It also assesses the impact of Parkinson's on specific dimensions of functioning and well-being. Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
Satisfaction and well-being visual analog scale | 16 weeks
  Patients will have to rate their feeling of satisfaction and well-being on a scale ranging from 0 (worst/lowest state of satisfaction and happiness) to 100 (highest state of satisfaction and happiness).

SECONDARY OUTCOMES:
MDS-Unified Parkinson Disease Rating Scale part III (MDSUPDRS) | 16 weeks
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive 50 question assessment of both motor and non-motor symptoms associated with Parkinson's. The investigators will administer part III only (motor examination). Higher scores reflect greater difficulties.
10-m walk test (10MWT) | 16 weeks
  This test is used and recommended as a measure of gait speed in Parkinson's disease (PD). It measures the speed in seconds of spontaneous and fastest rate walking.
Time up and go | 16 weeks
  At the signal from the assessor ("Go ahead"), the person should stand up and walk away.
  a comfortable and safe speed up to a line drawn on the floor (3 m further), turn, then come back and sit down. A first attempt should be made to familiarize the person with the test. The test therefore comprises an exercise and subsequently an "official" test. Results: the investigator starts the timing at "Go ahead" and stops it when the person has returned to a seated position.
  The time of the course (in seconds) is retained as the final score. The test will be judged positive (mobility disorders, risk of falling) if the score exceeds 12 to 14 seconds.
Montreal Cognitive Assessment (MoCA) | 16 weeks
  This scale includes 30 items assessing multiple cognitive domains: short-term memory (5 points); visuospatial abilities via clock drawing (3 points) and a cube copy task (1 point); executive functioning via an adaptation of Trail Making Test part B (1 point), phonemic fluency (1 point) and verbal abstraction (2 points); attention, concentration and working memory via target detection (1 point), serial subtraction (3 points), digits forward (1 point) and digits backward (1 point); language via confrontation naming with low-familiarity animals (3 points) and repetition of complex sentences (2 points); and orientation to time and place (6 points). Items are summed to create a score and the clinical cut-off score is equal to 26.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Site Ourthe-Amblève - CHU de Liège, Esneux, Liège
  - CNRF, Tinlot, Liège
  - CHU de Liège site Sart-Tilman, Liège

IPD SHARING:
Plan to Share IPD: No